CLINICAL TRIAL: NCT06137963
Title: Effectiveness of an Augmented Digital Diabetes Prevention Program for Adults With Prediabetes Having Elective Total Hip Arthroplasty: A Randomized Control Trial
Brief Title: Digital Diabetes Prevention Program Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is no longer feasible due to the increasing number of diabetic patients who are prescribed Ozempic and other GLP-1 agonists.
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-2194
Record Dates: First submitted 2023-09-14; First posted 2023-11-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-04

CONDITIONS: PreDiabetes
Keywords: prediabetes; hemoglobin a1c; hba1c; total hip arthroplasty
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: double-blind randomized control trial
Masking Description: Patient will be blinded because they will be told that they are getting the DPP within 0-6 months. RA's will not know what group patients are in because Transform10 will be asking all of the questionnaires via their platform.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transform10 Waitlist (Other): The control group will receive access to the Transform10 website at 6 months.
  Patients in this group will report their active minutes and weight via the Transform10 website throughout the 6 month-long programs. In addition, participants will take an Hba1c blood test at pre surgical screening, 6 months after their day of surgery and 1 year after their day of surgery as part of routine procedures.
  Interventions: Other: Transform10 Diabetes Prevention Program
- Transform10 (Experimental): Patients in this group will get access to the Transform10 website on their day of surgery.
  Patients in this group will report their active minutes and weight via the Transform10 website throughout the 6 month-long program. In addition, participants will have a repeat Hba1c test ordered at 6 months after their day of surgery and 1 year after their day of surgery as part of routine procedures.
  Interventions: Other: Transform10 Diabetes Prevention Program

INTERVENTIONS:
Other: Transform10 Diabetes Prevention Program — The Transform10 app includes a Centers for Disease Control (CDC)-approved diabetes prevention program.
  The self-paced curriculum and optional video content covers:
  * Strategies to overcome emotional eating using cognitive behavioral therapy principles.
  * Improving cardiovascular function with capacity-matched training programs using participants' estimated cardio scores.
  * An introductory-level course for increasing muscle and bone density foundation via strength training.
  * Education regarding physical therapy and expectations for patients.
  The Transform10 app also provides access to lifestyle coaches who discuss evidence-based information regarding hunger and insulin, macronutrient strategies, time-restricted intermittent fasting, and inflammation.

SUMMARY:
The aim of this study is to determine if completion of the Diabetes Prevention Program (DPP) via the Transform 10 website can significantly decrease hemoglobin A1c (HbA1c) levels and Body Mass Index (BMI) in prediabetic individuals undergoing total hip arthroplasty (THA) procedure.

As part of the standard procedure of the Centers for Disease Control (CDC)-approved DPP program, all study participants will report their active minutes and weight via the Transform10 website throughout the 6 month-long program. In addition, participants will have a repeat Hba1c test ordered at the end of the program by the medical director as part of routine procedures. The main questions it aims to answer are:

1. Is an augmented digital diabetes prevention program an effective strategy for weight loss in adults with prediabetes undergoing elective total hip arthroplasty?
2. Is an augmented digital diabetes prevention program an effective strategy to decrease HbA1c in adults with prediabetes undergoing elective total hip arthroplasty?
3. Is an augmented digital diabetes prevention program an effective strategy to improve postoperative outcomes and patient satisfaction in adults with prediabetes undergoing elective total hip arthroplasty?

Participants will be randomized to get the DPP on their day of surgery (intervention group) or get their DPP 6 months after their day of surgery (control group).

Comparing the intervention group to the control group, the researcher's primary outcome is change in percent of body weight before and after a 6-month intervention period.

DETAILED DESCRIPTION:
Glycemic, or blood sugar, control is an important factor associated with improved outcomes for patients after surgery. With one in three adults in the United States living with prediabetes, poor glycemic control has become an increasingly relevant indicator of postoperative complications. Glycemic control is commonly measured and referred to through the medical term hemoglobin A1c (HbA1c). Each percentage increase in HbA1c has been shown to be associated with increased complications around the time of surgery, intensive care unit admission, and hospital length of stay.

The aim of this study is to determine if completion of the Diabetes Prevention Program (DPP) via the Transform 10 website can significantly decrease HbA1c levels and Body Mass Index (BMI) in prediabetic individuals undergoing THA surgery. The main questions it aims to answer are:

1. Is an augmented digital diabetes prevention program an effective strategy for weight loss in adults with prediabetes undergoing elective total hip arthroplasty?
2. Is an augmented digital diabetes prevention program an effective strategy to decrease HbA1c in adults with prediabetes undergoing elective total hip arthroplasty?
3. Is an augmented digital diabetes prevention program an effective strategy to improve postoperative outcomes and patient satisfaction in adults with prediabetes undergoing elective total hip arthroplasty?

Participants will be randomized to get the DPP on their day of surgery (intervention group) or get their DPP 6 months after their day of surgery (control group).

Comparing the intervention group to the control group, the researcher's primary outcome is change in percent of body weight before and after a 6-month intervention period.

As part of the standard procedure of the Centers for Disease Control (CDC)-approved DPP program, all study participants will report their active minutes and weight via the Transform10 website throughout the 6 month-long program. In addition, participants will have a repeat Hba1c test ordered at the end of the program by the medical director as part of routine procedures.

The self-paced curriculum and optional video content covers:

* Strategies to overcome emotional eating using cognitive behavioral therapy principles.
* Improving cardiovascular function with capacity-matched training programs using participants' estimated cardio scores.
* An introductory-level course for increasing muscle and bone density foundation via strength training.
* Education regarding physical therapy and expectations for patients.

Participants will also have access to lifestyle coaches who discuss evidence-based information regarding hunger and insulin, macronutrient strategies, time-restricted intermittent fasting, and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Planned primary total hip arthroplasty for the indication of osteoarthritis at facility
* Age 18 - 64
* Overweight (BMI 25+ or 22+ if Asian)
* HbA1c 5.7%-6.4%
* Predicted ability to walk following procedure
* English or Spanish speaking
* Able to provide informed consent
* Willing to accept a random assignment
* Readiness for change
* ASA 1 or 2

Exclusion Criteria:

* Not meeting all inclusion criteria
* Diagnosed with Type I or II diabetes
* Diagnosed with congestive heart failure, coronary artery disease, chronic obstructive pulmonary disease, pulmonary hypertension
* Diagnosed with dementia or probable Alzheimer's disease
* Taking oral hypoglycemic agents other than Metformin
* Participating in a concurrent weight management program outside of HSS current protocol
* Unable to engage in walking as physical activity post-procedure
* Had bariatric surgery within the past 3 years or planning surgery within the next 12 months
* Anti-obesity or diabetes therapy within the preceding 4 months
* Any mental health condition, including eating disorders or alcohol/substance use, which would preclude full participation
* Self-report as currently pregnant or within 6 weeks of having given birth (or planning to become pregnant in the next 12 months)
* Unstable cardiac disease (i.e. heart attack/failure or stroke in the last 6 months, or currently in cardiac rehabilitation)
* On dialysis or an active organ transplant list
* Chronic kidney disease
* Untreated thyroid disease
* Cancer within the last 5 years unless skin cancer (i.e. currently or within the last 5 years in chemotherapy or radiation treatment)
* Unwilling to accept random assignment

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Change in percent of body weight before and after a 6 month intervention period. | Pre-surgical screening to 12 months post-operation
  body mass index will be measured at pre-surgical screening and again after a 6 month and 12-month period. The percent change in body weight will be recorded at program completion and at 6 months prior to program completion.

SECONDARY OUTCOMES:
Change in percent Hgb A1C after a 6 month intervention period. | Pre-surgical screening to 12 months post-operation
  hemoglobin a1c levels will be measured at pre-surgical screening and again after a 6 month and 12-month period. The percent change in hba1c level will be recorded.
Patient satisfaction. | 12 months post-operation
  Patient satisfaction will be a questionnaire that is asked by the Transform10 website 1 year after surgery. This questionnaire assesses how satisfied patients have been with their post operative pain management. This is reported on a scale from 0-10 with 0 being strongly dissatisfied and 10 being strongly satisfied.
Patient readiness assessment | day of surgery to 6 months prior to surgery
  Patients will be asked 8 questions upon access to the Transform10 program to assess their level of readiness for change. Each question asks if the patient is capable of a task and the responses range from "Sure I can", "Think I can", "Not sure I can", "Don't think I can".
Health related quality of life (HRQOL) | 12 months post-operation
  The health-related quality of life questionnaire will be asked via the transform10 website. This assesses how a patient's pain has impacted their day to day lives 12 months after their day of surgery. This is reported on a variety of scales depending on the questions asked. The scales include; 1 Excellent, 2 Very Good, 3 Good, 4 Fair, 5 Poor; 1 Much better now than one year ago, 2 Somewhat better now than one year ago, 3 About the same, 4 Somewhat worse now than one year ago, 5 Much worse now than one year ago; 1 Yes, limited a lot, 2 Yes, limited a little, 3 No, not limited at all; 1 Yes, 2 No; 1 Not at all, 2 Slightly, 3 Moderately, 4 Quite a bit, 5 Extremely; 1 None, 2 Very mild, 3 Mild, 4 Moderate, 5 Severe, 6 Very severe; 1 All of the time, 2 Most of the time, 3 A good bit of the time, 4 Some of the time, 5 A little of the time, 6 None of the time; 1 Definitely true, 2 Mostly true, 3 Don't know, 4 Mostly false, 5 Definitely false.
Possible postoperative complications | PACU arrival time to 12 months post-operation
  This will be recorded from Epic from post-operative care unit (PACU) admission to 12 months post-surgery.
Possible ICU Admission | PACU arrival time to 12 months post-operation
  This will be recorded from Epic from post-operative care unit (PACU) admission to 12 months post-surgery.
Possible patient readmission | PACU arrival time to 12 months post-operation
  This will be recorded from Epic from post-operative care unit (PACU) admission to 12 months post-surgery.
Postoperative length of stay | PACU arrival time to 12 months post-operation
  This will be recorded from Epic from post-operative care unit (PACU) admission to 12 months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jashvant Poeran, MD/PhD, Study Director — Hospital for Special Surgery, Department of Anesthesiology; Stephanie Cheng, MD, Principal Investigator — Hospital for Special Surgery, Department of Anesthesiology
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual patient data with other researchers.

REFERENCES:
- [Background] Couwenberg AM, de Beer FSA, Intven MPW, Burbach JPM, Smits AB, Consten ECJ, Schiphorst AHW, Wijffels NAT, de Roos MAJ, Hamaker ME, van Grevenstein WMU, Verkooijen HM. The impact of postoperative complications on health-related quality of life in older patients with rectal cancer; a prospective cohort study. J Geriatr Oncol. 2018 Mar;9(2):102-109. doi: 10.1016/j.jgo.2017.09.005. Epub 2017 Oct 10. PMID 29032962
- [Background] Santa Mina D, Scheede-Bergdahl C, Gillis C, Carli F. Optimization of surgical outcomes with prehabilitation. Appl Physiol Nutr Metab. 2015 Sep;40(9):966-9. doi: 10.1139/apnm-2015-0084. Epub 2015 May 13. PMID 26300015
- [Background] Wexler DJ, Nathan DM, Grant RW, Regan S, Van Leuvan AL, Cagliero E. Prevalence of elevated hemoglobin A1c among patients admitted to the hospital without a diagnosis of diabetes. J Clin Endocrinol Metab. 2008 Nov;93(11):4238-44. doi: 10.1210/jc.2008-1090. Epub 2008 Aug 12. PMID 18697862
- [Background] Flocke SA, Clark E, Antognoli E, Mason MJ, Lawson PJ, Smith S, Cohen DJ. Teachable moments for health behavior change and intermediate patient outcomes. Patient Educ Couns. 2014 Jul;96(1):43-9. doi: 10.1016/j.pec.2014.03.014. Epub 2014 May 1. PMID 24856449
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955
- [Background] Ackermann RT, O'Brien MJ. Evidence and Challenges for Translation and Population Impact of the Diabetes Prevention Program. Curr Diab Rep. 2020 Feb 20;20(3):9. doi: 10.1007/s11892-020-1293-4. PMID 32080770
- [Background] Kirley K, Sachdev N. Digital Health-Supported Lifestyle Change Programs to Prevent Type 2 Diabetes. Diabetes Spectr. 2018 Nov;31(4):303-309. doi: 10.2337/ds18-0019. PMID 30510384
- [Background] Cha E, Kim KH, Umpierrez G, Dawkins CR, Bello MK, Lerner HM, Narayan KM, Dunbar SB. A feasibility study to develop a diabetes prevention program for young adults with prediabetes by using digital platforms and a handheld device. Diabetes Educ. 2014 Sep-Oct;40(5):626-37. doi: 10.1177/0145721714539736. Epub 2014 Jun 20. PMID 24950683
- [Background] Wilson MG, Castro Sweet CM, Edge MD, Madero EN, McGuire M, Pilsmaker M, Carpenter D, Kirschner S. Evaluation of a Digital Behavioral Counseling Program for Reducing Risk Factors for Chronic Disease in a Workforce. J Occup Environ Med. 2017 Aug;59(8):e150-e155. doi: 10.1097/JOM.0000000000001091. PMID 28650899
- [Background] Michaelides A, Raby C, Wood M, Farr K, Toro-Ramos T. Weight loss efficacy of a novel mobile Diabetes Prevention Program delivery platform with human coaching. BMJ Open Diabetes Res Care. 2016 Sep 5;4(1):e000264. doi: 10.1136/bmjdrc-2016-000264. eCollection 2016. PMID 27651911

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT06137963/Prot_SAP_000.pdf